CLINICAL TRIAL: NCT05799105
Title: OPEN Versus InTact Capsule Proton Pump Inhibitors for the Treatment of Marginal Ulcers After Bariatric Surgery
Brief Title: OPEN Versus InTact Capsule Proton Pump Inhibitors for the Treatment of Marginal Ulcers
Acronym: OPEN-IT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Stephen Firkins (Other)
Responsible Party: Sponsor-Investigator, Stephen Firkins, Co-Director of Bariatric Endoscopy, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-024
Record Dates: First submitted 2023-02-28; First posted 2023-04-05 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-01

CONDITIONS: Marginal Ulcer
Keywords: marginal ulcer; bariatric surgery; gastric bypass; open capsule
MeSH Terms: conditions — Peptic Ulcer | interventions — Omeprazole

STUDY DESIGN:
Intervention Model Description: prospective single-blinded randomized control trial
Who Masked: Care Provider, Investigator
Masking Description: Endoscopists diagnosing and surveying healing of marginal ulcers will be blinded to the subject's treatment arm. A single, unmasked provider will be responsible for randomizing and prescribing either open- or intact-capsule PPI after subjects are enrolled in the study. This unmasked provider will not take part in diagnosis, monitoring or assessment of ulcer healing, or in data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Open-capsule (Experimental): Subjects in this arm will be treated with omeprazole 40 milligrams twice daily (or alternative medication if not covered by the subject's insurance) taken as an open-capsule until confirmed ulcer healing.
  Interventions: Drug: Omeprazole 40 milligrams
- Intact-capsule (Active Comparator): Subjects in this arm will be treated with omeprazole 40 milligrams twice daily (or alternative medication if not covered by the subject's insurance) taken as an intact-capsule until confirmed ulcer healing or potential cross-over.
  Interventions: Drug: Omeprazole 40 milligrams

INTERVENTIONS:
Drug: Omeprazole 40 milligrams — Subjects will be randomized to treatment with either open-capsule or intact-capsule omeprazole to assess effect on ulcer healing times. If interim analysis illustrates significantly improved healing in the open-capsule group, the control (intact-capsule) arm will be allowed to cross-over to open-capsule and be followed until confirmed ulcer healing.
  Other Names: Prilosec; Losec

SUMMARY:
The goal of this clinical trial is to identify the most effective way to take acid-blocking medications to treat stomach ulcers in patients who have undergone gastric bypass surgery. The main questions it aims to answer are:

* is taking an acid-blocking medication by opening the capsule and only taking the contents of the capsule (open-capsule) more or less effective than taking the capsule as a whole (intact-capsule) for treating ulcers in patients who have a history of gastric bypass surgery?
* does taking the open versus intact medication decrease the number of procedures and complications from untreated ulcers?

Participants with ulcers will be instructed to take acid-blocking medications (called proton-pump inhibitors) either by opening the capsule and taking only the contents or by taking the capsule whole. These medications are the gold standard for treatment of stomach ulcers. Participants will be asked to undergo an upper endoscopy (EGD) every 3 months to monitor the healing of the ulcers.

Researchers will compare how quickly the ulcers heal depending on which way the medications are taken (opened up or as a whole).

DETAILED DESCRIPTION:
Marginal ulcers (ulcers formed at the surgery site between the stomach and the intestines) are a common complication of bariatric surgery, ranging in frequency from 0.6-25% of patients. Furthermore, roughly 17% of patients with marginal ulcers require repeat procedures or surgery for severe complications such as bleeding, perforation, stricture, and fistulas.

Proton pump inhibitors (PPIs), which act by block acid secretion from the stomach, are the gold standard for treatment of ulcers. There is limited data showing that opening the PPI capsule and taking only the contents greatly improves healing of marginal ulcers after gastric bypass surgery. This is likely due to the much smaller stomach, faster passage through the stomach and decreased ability of the intact PPI medication to be broken down and absorbed.

This would be the first clinical trial to confirm whether this is true, which would support all patients who get ulcers after gastric bypass surgery to be treated with open-capsule PPI medications.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with marginal ulceration post-gastric bypass on upper endoscopy

Exclusion Criteria:

* Refusal to start PPI medication OR current open-capsule PPI use at the time of diagnosis of the marginal ulcer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2025-12-23 (Estimated); Study Completion 2025-12-23 (Estimated)

PRIMARY OUTCOMES:
Ulcer healing | On average, 3 months to 12 months
  Rate of ulcer healing in each treatment arm, defined as resolution of previously-seen ulcer on upper endoscopy

SECONDARY OUTCOMES:
Ulcer healing time | On average, 3 months to 12 months
  Time to ulcer healing, defined as (date of ulcer healing) - (date of ulcer diagnosis)
pH of gastric pouch | Upon initial enrollment endoscopy
  pH of the gastric pouch fluid will be obtained during initial endoscopy and tested with litmus paper. pH data will be compared between the two treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Firkins, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

REFERENCES:
- [Background] English WJ, DeMaria EJ, Hutter MM, Kothari SN, Mattar SG, Brethauer SA, Morton JM. American Society for Metabolic and Bariatric Surgery 2018 estimate of metabolic and bariatric procedures performed in the United States. Surg Obes Relat Dis. 2020 Apr;16(4):457-463. doi: 10.1016/j.soard.2019.12.022. Epub 2020 Jan 3. PMID 32029370
- [Background] Coblijn UK, Goucham AB, Lagarde SM, Kuiken SD, van Wagensveld BA. Development of ulcer disease after Roux-en-Y gastric bypass, incidence, risk factors, and patient presentation: a systematic review. Obes Surg. 2014 Feb;24(2):299-309. doi: 10.1007/s11695-013-1118-5. PMID 24234733
- [Background] Ribeiro-Parenti L, Arapis K, Chosidow D, Marmuse JP. Comparison of marginal ulcer rates between antecolic and retrocolic laparoscopic Roux-en-Y gastric bypass. Obes Surg. 2015 Feb;25(2):215-21. doi: 10.1007/s11695-014-1392-x. PMID 25085224
- [Background] Pyke O, Yang J, Cohn T, Yin D, Docimo S, Talamini MA, Bates AT, Pryor A, Spaniolas K. Marginal ulcer continues to be a major source of morbidity over time following gastric bypass. Surg Endosc. 2019 Oct;33(10):3451-3456. doi: 10.1007/s00464-018-06618-5. Epub 2018 Dec 12. PMID 30543040
- [Background] Di Palma A, Liu B, Maeda A, Anvari M, Jackson T, Okrainec A. Marginal ulceration following Roux-en-Y gastric bypass: risk factors for ulcer development, recurrence and need for revisional surgery. Surg Endosc. 2021 May;35(5):2347-2353. doi: 10.1007/s00464-020-07650-0. Epub 2020 May 18. PMID 32424625
- [Background] Tansel A, Graham DY. New Insight Into an Effective Treatment of Marginal Ulceration After Roux-en-Y Gastric Bypass. Clin Gastroenterol Hepatol. 2017 Apr;15(4):501-503. doi: 10.1016/j.cgh.2016.12.025. Epub 2017 Jan 3. No abstract available. PMID 28062217
- [Background] Schulman AR, Chan WW, Devery A, Ryan MB, Thompson CC. Opened Proton Pump Inhibitor Capsules Reduce Time to Healing Compared With Intact Capsules for Marginal Ulceration Following Roux-en-Y Gastric Bypass. Clin Gastroenterol Hepatol. 2017 Apr;15(4):494-500.e1. doi: 10.1016/j.cgh.2016.10.015. Epub 2016 Oct 20. PMID 27773764

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-09): https://cdn.clinicaltrials.gov/large-docs/05/NCT05799105/Prot_SAP_000.pdf